CLINICAL TRIAL: NCT01640912
Title: A Phase 1 Single Center, Randomized, Double-Blind, Ascending Dose, Within-Subject Controlled Study of RXI-109 for the Treatment of Incision Scars Made in the Pannus of Healthy Women Who Will Later Undergo Elective Abdominoplasty
Brief Title: Evaluation of the Safety, Pharmacokinetics, and Preliminary Effect on Scar Formation by RXI-109
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RXi Pharmaceuticals, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RXI-109-1201
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Cicatrix; Scar Prevention
Keywords: Scar; Scar prevention; Fibrosis
MeSH Terms: conditions — Cicatrix; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RXI-109 (Experimental)
  Interventions: Drug: RXI-109
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RXI-109 — Single intradermal injection of RXI-109 at incision sites
  Arms: RXI-109
Drug: Placebo — Single intradermal injection of placebo at incision sites
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of a single intradermal administration of RXI-109 at small surgical incisions in the abdominal skin that will later be removed during an elective abdominoplasty. The effect of RXI-109 versus placebo on scarring at these incision sites will be evaluated visually and histologically.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a female in general good health with normal screening values
* Subject must be a good surgical candidate for an elective abdominoplasty
* Subjects must not be pregnant or lactating and utilize an effective method of contraception (if child-bearing potential exists)

Exclusion Criteria:

* Currently pregnant or lactating
* BMI greater than 35 at screening
* Use of tobacco or nicotine-containing products within the month prior to enrollment and while on study
* Any medical condition or current therapy which would make the subject unsuitable for this study in the opinion of the PI

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of intradermal administration of RXI-109 | 12 weeks
  Evaluate safety and tolerability of RXI-109 at site of intradermal injection. Examination and assessment of any and all local and systemic toxicities

SECONDARY OUTCOMES:
To assess the effect of RXI-109 on scar formation following small surgical incisions | 12 weeks
  Visual outcome and histology of scars will be assessed. Digital images of the RXI-109 and placebo-treated incisions/scars will be captured and assessed by a masked, independent, expert panel.

CONTACTS AND LOCATIONS:
Locations (1):
- St Louis, Missouri, United States